CLINICAL TRIAL: NCT01999101
Title: A Safety Pilot Study of Px-104 in Non-alcoholic Fatty Liver Disease (NAFLD) Patients
Brief Title: Safety Pilot Study of Farnesoid X Receptor (FXR) Agonist in Non-alcoholic Fatty Liver Disease (NAFLD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phenex Pharmaceuticals AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHS-Px-104-II-01
Record Dates: First submitted 2013-11-19; First posted 2013-12-03 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2014-11

CONDITIONS: Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Px-104 (Experimental): Px-104 capsules, 5 mg
  Interventions: Drug: Px-104

INTERVENTIONS:
Drug: Px-104 — 28 days treatment

SUMMARY:
The primary aim of the study is to evaluate the safety and tolerability of Px-104 in NAFLD patients and to assess the influence of Px-104 on hepatic fat.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD patients
* Weight > 65 kg
* BMI > 25 and < 40
* Negative blood or urine pregnancy test (for females of childbearing potential) collected at screening followed by another negative serum pregnancy test collected within 24 hours prior to the first dose of study drug.
* Contraception: Female patients must be postmenopausal, surgically sterile, or if premenopausal, must be prepared to use at least two effective (≤1% failure rate) method of contraception during the course of the study and for 14 days after the end of dosing. Male patients with female partners of child bearing potential must be prepared to use at least two effective methods of contraception with all sexual partners unless they have had a prior vasectomy
* Must be willing and able to give written informed consent and agree to comply with the study protocol.
* Sinus rhythm in 12-lead ECG

Exclusion Criteria:

* Evidence of excessive alcohol, drug or substance abuse (excluding marijuana use) within 1 year of first dose.
* History or other evidence of a medical condition associated with chronic liver disease other than.
* History or other evidence of decompensated liver disease (Child-Pugh Grade B or higher), coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites, hepatic encephalopathy, and bleeding from esophageal varices are conditions consistent with decompensated liver disease.
* Concomitant intake of fibrates or statins (at least 4-6 weeks before start; considering half life of medication).
* Any clinically relevant findings in ECG (identified via 24h-Holter ECG or 12-Lead ECG) at screening
* History of any structural cardiac disease.
* In addition, patients with documented or presumed unstable coronary artery disease, stable or unstable cardiovascular disease or cerebrovascular disease.
* One or more of the following conditions: (1) poorly controlled hypertension, OR (2) screening or baseline blood pressure ≥ 160 mmHg for systolic OR (3) screening or baseline blood pressure ≥ 100 mmHg for diastolic blood pressure.
* Type I or II diabetes with HbA1C > 6.5% at screening and/or fasting plasma glucose > 7mmol/L (> 126 mg/dl).
* History or other evidence of a clinically relevant ophthalmologic disorder due to diabetes mellitus or hypertension or history or other evidence of severe retinopathy (e.g., cytomegalovirus, macular degeneration).
* Known sensibility to any ingredients contained in the investigational medicinal product (IMP)
* All conditions that do not allow magentic resonance (MR) assessments
* History of having received any investigational drug ≤ 3 months and/or 6 x half-life prior to the first dose of study drug or the expectation that such drugs will be used during the study. Patients enrolled in this study cannot be enrolled in another study for either research, diagnostic or treatment purposes.
* Woman with childbearing potential unless using adequate contraception (see inclusion criteria); females who are pregnant or breast feeding.
* History of severe allergic
* Evidence of an active or suspected cancer, or a history of malignancy within the last 2 years, with the exception of patients with basal cell carcinoma that has been excised and cured.
* History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* History of bleeding disorders or anticoagulant use
* History or other evidence of chronic pulmonary disease associated with functional limitation.
* History of uncontrolled severe seizure disorder.
* Poorly controlled thyroid dysfunction.
* History of major organ transplantation with an existing functional graft.
* Any signs of acute infection or inflammation
* History or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study.
* Any herbal supplements containing silymarin, tocopherol, vitamin C, riboflavins, proflavins, curcumin. (at least 4-6 months before the study)
* Positive test at screening for anti-Hepatits A virus (HAV) Immunoglobulin M (IgM), Hebatitis B surface antigen (HBsAg), Anti-Hepatits B core Antigen Immunglobulin M antibody (anti-HBc IgM Ab), or anti-HIV Ab.
* Subjects who have undergone surgery within the last 3 months.
* Subjects who have had a prior gastrointestinal surgery.
* Subjects who will be unavailable for the duration of the trial, who are unlikely to be compliant with the protocol, or who are felt to b unsuitable by the investigator for any other reason
* Imprisonment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety | 28 days
  Analysis of clinical chemistry, hematology, and assessment of clinical signs and adverse events over 28 days. Change day 28 vs. day 1

SECONDARY OUTCOMES:
Change of hepatocellular lipid content | day 1 and day 28
  Measurement of hepatic fat (%) by Magnetic resonance spectroscopy (MRS), change day 28 vs. day 1
Changes in oral glucose tolerance test (oGTT) | baseline and day 27
  Measurement of plasma glucose level (mg/dL)
Change from baseline in fibroblast growth factor 19 (FGF-19) | days 1, 7, 14, 21 and 28
  Measurement by ELISA (pg/mL)
Change from baseline in plasma bile acid concentration | days 1, 7, 14, 21, and 28.
  Assessment by LC-MS/MS (µmol/L)
Pharmacokinetics of Px-104 and conjugates | day 1 and day 28
  Measurement by LC-MS/MS (ng/mL). AUC, Cmax and other pk parameters

OTHER OUTCOMES:
Changes in the Saccharose-Lactulose-Mannitol + Sucralose (SLM+S) Test to evaluate the intestinal permeability | baseline and day 27
  Measurement of urinary concentrations of Saccharose, Lactulose, Mannitol and Sucralose by HPLC
Assessment of liver steatosis by CAP-Fibroscan | baseline and day 28
  Measurement of hepatic fat (%) by CAP-Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, Professor Dr med, Principal Investigator — Medical University Vienna
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine III, Vienna, Austria